CLINICAL TRIAL: NCT02584907
Title: Effect of Fat Based Versus Glucose Based Enteral Nutrition on Serum Glucose Levels and Clinical Outcome in Hyperglycemic Patients in ICU
Brief Title: Fat Based Enteral Nutrition for Blood Glucose Control in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Assistant Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1395/34199
Record Dates: First submitted 2015-10-19; First posted 2015-10-23 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Hyperglycemia
Keywords: Critically ill; Diet; Blood glucose
MeSH Terms: conditions — Hyperglycemia; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Fat Enteral Nutrition (Experimental): Diet in high fat group will be 20% from protein, 45% from fat and 35% from carbohydrate
  Interventions: Other: High Fat Enteral Nutrition
- Standered Enteral Nutrition (No Intervention): Diet in standard group will be 20% from protein, 30% from fat and 50% from carbohydrate

INTERVENTIONS:
Other: High Fat Enteral Nutrition — Diet in high fat group will be 20% from protein, 45% from fat and 35% from carbohydrate
  Arms: High Fat Enteral Nutrition

SUMMARY:
In this randomized, double-blind clinical trial, eligible hospitalized ICU patients with EN will be included. Patients will be divided into two groups. The control group with the standard EN and intervention group with high fat EN. 50% of the total fat will be provided by olive oil. Nutritional intake record form will be completed and daily calorie intake will be calculated. High fat EN feeding will be offered for 15 consecutive days maximally. At the end of the study mean blood glucose, duration of hospitalization and rate of infection will be compared in two groups.

DETAILED DESCRIPTION:
In this randomized, double-blind clinical trial, 88 eligible hospitalized ICU patients with EN will be included. Written consent form will be completed. Physical examination will be done by specialist and nutritional care process will be offered by an RD. Demographic, laboratory and nutritional data will be extracted and entered in prepared form. Venous blood samples will be taken and laboratory values will be measured and recorded at specified times. Patients will be divided into two groups. The control group with the standard EN (Protein; 20% carbohydrate; 50% and fat; 30% from total calories) and intervention group with high fat EN (Protein; 20% carbohydrate; 35% and fat; 45% from total calories). 50% of the total fat will be provided by olive oil. Any feeding rout such as naso - gastric , Percutaneous endoscopic gastrostomy (PEG ) or Percutaneous endoscopic jejunostomy (PEJ) with Intermittent feeding protocol will be accepted feeding method . Nutritional intake record form will be completed and daily calorie intake will be calculated. High fat EN feeding will be offered for 15 consecutive days maximally

ELIGIBILITY:
Inclusion Criteria:

* Being on Enteral Nutrition
* BS≥ 200mg/dl
* Without Renal and Liver Failure
* Without Hyperlipidemia and Nephrotic Syndrome
* Without Infection
* Without Obesity

Exclusion Criteria:

* Death or Discharge before Day 7

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 1 year

SECONDARY OUTCOMES:
Length of Stay in ICU | 1 year
Occurrence of Infection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, Ph.D, Study Chair — Faculty of Nutrition and Food Sciencees, Shahid Beheshti University of Medical Sciences
Locations (1):
- Faculty of Nutrition Sciences and Food Technology, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wewalka M, Drolz A, Zauner C. Influence of fat-based versus glucose-based enteral nutrition formulas on glucose homeostasis. Crit Care. 2013; 17(Suppl 2): P250. Published online 2013 Mar 19. doi: 10.1186/cc12188. PMCID: PMC3642614.
- See also: Critical Care — http://www.ccforum.com